CLINICAL TRIAL: NCT01497912
Title: Treatment Effects of Atorvastatin on Hemostasis and Skin Microcirculation in Patients With Type 1 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Dnr 04-681/2; Dnr 151:2004/52378 (Other: Swedish Medical Products Agency)
Record Dates: First submitted 2011-12-22; First posted 2011-12-23 (Estimated); Last update posted 2011-12-23 (Estimated); Status verified 2005-01

CONDITIONS: Type 1 Diabetes Mellitus; Dyslipidemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Dyslipidemias | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin (Active Comparator): Atorvastatin 80mg once daily
  Interventions: Drug: Atorvastatin
- Placebo (Placebo Comparator): Matched placebo tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin 80mg once daily for 8 weeks
  Arms: Atorvastatin
Drug: Placebo — Placebo tablet once daily for 8 weeks
  Arms: Placebo

SUMMARY:
Patients with type 1 diabetes are at increased risk of vascular complications both in the micro- and macrocirculation. Hyperglycemia plays a major role in the development of these vascular complications, but other factors such increased platelet adhesion and aggregation, elevated levels of plasma fibrinogen, altered fibrin network structure, increased thrombin generation, dyslipidemia and endothelial dysfunction may contribute.

Lipid-lowering therapy with statins is effective in prevention of cardiovascular events in individuals at increased risk. Statins seem to exert beneficial effects on hemostasis and vasculature that are independent of their lipid-lowering properties.

The aim of the present study was to investigated the effects of intensive LDL-cholesterol-lowering therapy with atorvastatin on fibrin network permeability (primary variable) and other aspects of hemostasis in patients with type 1 diabetes and dyslipidemia. Furthermore, the effects of atorvastatin therapy on skin microvascular function was also investigated.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes
* level of plasma LDL-cholesterol >2.5mmol/L and/or total cholesterol >4.5mmol/L

Exclusion Criteria:

* History of macrovascular events

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-01; Primary Completion 2009-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Fibrin network permeability | 8 weeks

SECONDARY OUTCOMES:
platelet and endothelial microparticles | 8 weeks
skin microvascular reactivity | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Department of Clinical Sciences, Danderyd Hospital, Stockholm, Sweden

REFERENCES:
- See also: PubMed — http://www.ncbi.nlm.nih.gov/pubmed/20637495